CLINICAL TRIAL: NCT07336667
Title: 족저압 요약 피드백 제공 유무에 따른 로봇보조보행훈련의 효과: 편마비 환자의 보행 대칭성과 균형에 미치는 영향; The Effect of Robot-Assisted Gait Training With or Without Plantar Pressure Summary Feedback: Impact on Gait Symmetry and Balance in Hemiplegic Patients
Brief Title: The Effect of Robot-Assisted Gait Training With or Without Plantar Pressure Summary Feedback: Impact on Gait Symmetry and Balance in Hemiplegic Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yeonji Choi (Other)
Responsible Party: Sponsor-Investigator, Yeonji Choi, researcher, Sahmyook University
Organization: Sahmyook University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-08-026-003
Record Dates: First submitted 2025-12-11; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Hemiplegia
Keywords: Chronic hemiplegic stroke; robot assisted gait training; Lokomat; GaitRite; Plantar pressure feedback
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lokomat with plantar pressure summary feedback (Experimental): Participants receive 30 minute Lokomat(robot-assisted gait training) with real-time feedback plus additional plantar pressure summary feedback. Training is provided 3 times per week for 4 weeks. Balance and gait symmetry are assessed before and after the intervention
  Interventions: Device: Lokomat robot assisted gait training; Other: Plantar pressure summary feedback
- Real-time feedback(biofeedback program) (Active Comparator): Participants receive 30 minute Lokomat(robot-assisted gait training) training with real-time feedback only. Training is provided 3 times per week for 4 weeks. Balance and gait symmetry are assessed before and after the intervention.
  Interventions: Device: Lokomat robot assisted gait training

INTERVENTIONS:
Device: Lokomat robot assisted gait training — Lokomat robot assisted gait training for 30 minutes per session, 3 times per week, for 4 weeks. Real-time(biofeedback graph) visual and auditory feedback provided by the Lokomat system is used during gait training in both groups.
Other: Plantar pressure summary feedback — Experimental group, plantar pressure data are collected during each Lokomat session using instrumented insoles. After each session, session by session plantar pressure summary feed back and gait symmetry is provided to the participant to promote more symmetrical gait. The control group does not receive this plantar summary feedback.
  Arms: Lokomat with plantar pressure summary feedback

SUMMARY:
The goal of this randomized, single-blind clinical trial is to learn whether a 4-week Lokomat-based gait training program with plantar pressure feedback can improve gait symmetry and balance in adult patients with chronic hemiplegic stroke. The main questions it aims to answer are:

Does Lokomat training with plantar pressure feedback improve spatiotemporal gait symmetry, as measured with the GAITRite system, more than Lokomat training without plantar pressure feedback? Does this intervention lead to greater improvements in balance and walking speed, assessed by the Berg Balance Scale (BBS) and the 10-Meter Walk Test (10MWT), compared with conventional Lokomat training? Researchers will compare a group receiving Lokomat training with both real-time feedback and additional summary plantar pressure feedback to a group receiving Lokomat training with real-time feedback only, to see if adding plantar pressure feedback results in superior gains in gait symmetry, balance, and walking ability.

Participants will be adult inpatients with chronic hemiplegic stroke. They will be randomly assigned to one of the two training groups and will receive Lokomat-based gait training three times per week for 30 minutes per session over four weeks. Before and after the intervention period, participants will undergo gait analysis using the GAITRite walkway and clinical assessments including the BBS and 10MWT.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with hemiplegia after stroke who are currently admitted to or visiting the rehabilitation therapy department of Seoul Brain Hospital in Yeongdeungpo-gu, Seoul, Republic of Korea.
* Chronic stage after stroke onset of at least 6 months.
* Diagnosis of unilateral hemiplegia.
* Mini-Mental State Examination(MMSE) score ≥ 24, with ability to understand the study procedures and provide informed consent.
* Functional Ambulation Catefories(FAC) score of 1-2(FAC 0 excluded.)
* Ability to communicate voluntarily for participation and consent.
* Suiable physical condition for robot-assisted gait training(RAGT) and use of Lokomat device, including body weight ≤ 135 kg and height between approximately 150 cm and 2.0 m.

Exclusion Criteria:

* MMSE score ≤ 23, indicating difficulty understanding the study procedures or expressing informed consent.
* History of major psychiatric disorders such as schizophrenia, major depressive disorder, or bipolar disorder.
* Uncontrolled cardiovascular or respiratory disease that makes gait training unsafe, such as uncontrolled hypertension, significant arrhythmia, angina, or acute exacerbation of respiratory disease.
* Orthopedic or neuromuscular conditions that prevent safe robotic gait training, including:
* Lower limb surgery or fracture within the previous 3 months.
* Moderate-to-severe joint contracture or severe spasticity (e.g., Modified Ashworth Scale ≥ 3).
* Clinically significant leg-length discrepancy (≥ 2 cm).
* Severe skin infection, pressure ulcer, or other skin condition at the harness or strap contact areas that makes physical contact difficult.
* Low back pain, dizziness, orthostatic hypotension, or other symptoms that prevent continuation of RAGT.
* Acute or recurrent neurological events within the previous 3 months (e.g., recurrent cerebrovascular events).
* Any other medical condition that the principal investigator judges to make participation unsafe.

Vulnerable Populations:

This study includes only adult participants and does not enroll legally vulnerable populations such as minors or pregnant women. For inpatients, potential reduction in voluntariness due to relationships with treating clinicians is minimized by obtaining consent from a non-treating researcher, allowing sufficient time for decision-making, permitting withdrawal at any time without penalty, and allowing a caregiver to be present during the consent process if desired.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Change in gait symmetry(GaitRite) | Change from baseline to 4 weeks after randomization(end of intervention)
Change in gait symmetry(10-meter walk test) | Change from baseline to 4 weeks after randomization(end of intervention)

SECONDARY OUTCOMES:
Change in balance performance(Berg Balance Test) | Change from baseline to 4 weeks after randomization(end of intervention)
Change in balance performance(Timed Up and Go test) | Change from baseline to 4 weeks after randomization(end of intervention)

CONTACTS AND LOCATIONS:
Overall Officials: seongwon Lee, PhD, PT, Principal Investigator — Sahmyook University, Department of Physical Therapy
Locations (1):
- Duksoo Medical Foundation Seoul Brain Hospital, Seoul, Seoul, South Korea